CLINICAL TRIAL: NCT03028454
Title: Effects of Ginger on Muscle Soreness and Dysfunction Stemming From Downhill Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Assistant Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 934537-3
Record Dates: First submitted 2017-01-14; First posted 2017-01-23 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginger Root Capsule (Experimental)
  Interventions: Dietary Supplement: Ginger Root
- Placebo Capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger Root — Capsules containing 250 mg of ginger root extract standardized to contain at least 5% gingerol compounds, as well as an additional 225 mg of regular ginger root.
  Arms: Ginger Root Capsule
Dietary Supplement: Placebo — Capsules containing rice flour powder.
  Arms: Placebo Capsule

SUMMARY:
The objective of the study is to determine whether five days of ginger (Zingiber officinale) supplementation is effective at reducing muscle soreness and improving muscle function following downhill running. Long-distance running is often associated with acute muscle pain, swelling, and reduced muscle functioning, and consequently, many runners utilize non-steroidal anti-inflammatory drugs (NSAID). NSAID use is associated with gastrointestinal side-effects such as stomach discomfort, nausea, dyspepsia, asymptomatic ulcers, and symptomatic ulcers that, although rare, can be fatal. Ginger is a botanical compound that is Generally Recognized as Safe by the Food and Drug Administration (FDA). Evidence from osteoarthritis, dysmenorrhea, and resistance-training models indicate that ginger is effective at reducing general pain and muscle soreness. Therefore, this study will supplement 60 runners with roughly 1.5 g/day of ginger root or a placebo for 2 days prior to, the day of, and 2 days after downhill running. Participants will be evaluated for muscle soreness and function before and after the downhill run.

ELIGIBILITY:
Inclusion Criteria:

* Be currently running ≥10 miles per week
* Have completed at least one run >40 minutes over the past month

Exclusion Criteria:

* Have no allergies to ginger
* Willing to avoid pain-relieving medications for the duration of the study
* Have no history of bleeding disorders nor currently taking blood thinners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Muscle Soreness Change | Two days before a 40-minute downhill run, the day of a 40-minute downhill run, 24 hours after a 40-minute downhill run and the two days after a 40-minute downhill run
  Participants will be asked to mark a slash on a 100 mm line the muscle soreness of their lower extremities, with descriptors of "no soreness'' indicated at 0 and ''unbearably painful" at 100. Participants will rate overall lower-extremity soreness at rest, while performing a stand-to-sit movement, and while running at a moderate pace.

SECONDARY OUTCOMES:
Pain Pressure Threshold Change | Two days before a 40-minute downhill run, the day of a 40-minute downhill run, and two days after a 40-minute downhill run
  An algometer will be applied to the participant's quadriceps muscle. An algometer is a handheld device with an integral load cell that transduces the pressure applied to the participant. The investigator will apply force slowly and smoothly while the participant concentrates on when the force applied by the investigator transitions from a feeling of pressure to a feeling of pain. The force level applied when the participant begins to feel pain will be considered the pain pressure threshold. The location of the measurement will be 10 cm above the superior crest of the patella. The average of two measurements will be taken.
Vertical Jump Test Change | Two days before a 40-minute downhill run, the day of a 40-minute downhill run, and two days after a 40-minute downhill run
  Participants will jump as high as possible using the squat jump technique. Participants will perform three trials.
1.5-mile Run Change | Two days before a 40-minute downhill run and two days after a 40-minute downhill run
  Participants will complete a maximal effort 1.5-mile run on a motorized treadmill.
Lung Function Change | Two days before a 40-minute downhill run and two days after a 40-minute downhill run
  Participants' lung function will be tested before the 1.5-mile run and at 1, 5, 10, 15, and 20 minutes post-exercise. Lung function will be assessed with a spirometer by having participants perform a maximal forced expiration. Breathing difficulty will also be measured before and after the run with the Modified Borg Dyspnea Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States